CLINICAL TRIAL: NCT00548704
Title: A Clinical Trial on Topotect® (Dexrazoxane) in the Treatment of Accidental Extravasation of Anthracycline Anti-cancer Agents
Brief Title: A Clinical Trial on Topotect® (Dexrazoxane) in the Treatment of Accidental Extravasation of Anthracyclines
Status: Completed | Phase: Phase 2 / Phase 3 | Type: Interventional
Sponsor: Valerio Therapeutics (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: TT02
Record Dates: First submitted 2007-10-23; First posted 2007-10-24 (Estimated); Last update posted 2015-10-21 (Estimated); Status verified 2013-11

CONDITIONS: Extravasation
Keywords: Extravasation; Anthracyclines
MeSH Terms: interventions — Dexrazoxane; Razoxane

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Drug: Dexrazoxane
  Other Names: Totect

SUMMARY:
The purpose of this study is

* To prevent progression of a lesion caused by anthracycline extravasation into necrosis, which would require surgical intervention
* To prevent development of deep tissue necrosis and destruction leading to impaired limb function and neurological deficit
* To prevent postponement of the scheduled cancer treatment due to the treatment of the extravasation

DETAILED DESCRIPTION:
Accidental extravasation of anthracyclines, e.g. doxorubicin and its derivative epirubicin, may cause progressive tissue destruction including serious damage of the skin, the subcutaneous tissue, muscles, and nerves.

The patient may suffer from acute local symptoms such as pain and swelling, which may progress into blistering and necrosis. Subsequently dysesthesia, skin atrophy, disfigurement, and impaired limb function may be the consequence.

Surgical removal of all affected tissue is required and the debridement often necessitates split skin grafting. The patient is thus subjected to the distress of major surgery, which in turn leads to delay of further cytotoxic treatment.

Preclinical animal studies as well as a clinical multicenter phase II trial have demonstrated a highly significant efficacy of dexrazoxane in preventing tissue destruction caused by anthracyclines.

This confirmatory trial will determine the effect of Topotect® (dexrazoxane) as an acute antidote in patients with anthracycline extravasation.

Orphan drug status TopoTarget A/S was granted designation for Topotect® as an orphan medical product for the treatment of anthracycline extravasations by the European Commission in September 2001 and by the FDA in ???.

Purpose

Primary objectives:

• To prevent progression of the anthracycline extravasation lesion as tissue ulceration and necrosis requiring surgical intervention

Secondary objectives:

* To prevent development of deep tissue necrosis and destruction leading to late sequelae as impaired limb function and neurological deficit
* To prevent postponement of the scheduled cancer treatment due to the treatment of the extravasation
* To evaluate the tolerance to and/or toxicity of Topotect® used for this indication, according to the indicated schedule

Trial design This is an open-label, non-randomised phase II/III trial. Thirty -five evaluable patients with anthracycline extravasations will be treated.

Extravasation is determined by the presence of pain, and/or swelling, and/or redness at the site where anthracycline leakage is suspected to have occurred. The extravasations are subsequently confirmed in each patient by fluorescence microscopy of at least two punch biopsies at the time of the accident.

Success criteria The prevention of surgical intervention, necrosis and late sequelae evaluated 3 months after the extravasation.

Safety features

* Toxicity caused by Topotect® will be examined by haematology and blood chemistry, questions are asked on any discomfort. Scheduled clinical examinations are performed
* A systematic clinical evaluation of the marked area of skin covering the area of extravasation will be performed in order to evaluate the need for surgery
* Sequential colour photographs of the involved skin will be taken

Medical Treatment Patients are treated with intravenous infusion of Topotect® administered once daily on three consecutive days at the following doses: 1,000 mg/m2 + 1,000 mg/m2 + 500 mg/m2. The first dose is administered as soon as possible and within 6 hours of the extravasation and the next two doses at 24 and 48 hours after the first infusion.

ELIGIBILITY:
Inclusion Criteria:

1. All cancer patients treated with anthracyclines
2. Informed consent must be obtained from the patient
3. Patients suspected to have been exposed to extravasation (leakage) of anthracycline, defined as:

   1. A primary assessment by the physician on duty, which would activate the standard departmental procedure for treatment of anthracycline extravasation.
   2. The presence of at least one of the following symptoms: pain, swelling or redness at the site where the anthracycline leakage is suspected to have occurred.
4. Suspicion of anthracycline extravasation from a central venous access device
5. The Topotect® infusion must be started < 6 hours after the accident
6. 18 years of age or older
7. Performance status (PS) < 2

Exclusion Criteria:

1. Known allergy towards dexrazoxane
2. Reasonable suspicion of extravasation by other compounds than anthracyclines through the same intravenous access, e.g. vincristine, mitomycin, and vinorelbine, all of which may cause ulceration
3. AST (aspartate aminotransferase) or ALT (alanine aminotransferase), bilirubin, LDH (lactate dehydrogenase), alkaline phosphatase >3 x upper normal value
4. Neutrophils CTC (common toxicity criteria) ≥ grade 2. (neutrophils 1.5 x 109/L, ≥1,500/mm3)
5. Platelets CTC ≥ grade 2. (platelets ≥75.0 x 109/L, <75,000/mm3).
6. Topical use of DMSO (dimethylsulfoxide) at the area of the accident
7. Administration of dexrazoxane within the last 3 weeks
8. Pregnant or nursing women
9. Women of childbearing age and potential, who do not use an efficient contraceptive (e.g. the Pill or a diaphragm plus a spermicide) for at least 3 months prior to the start of trial medication

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 57 (Actual)
Dates: Start 2002-04; Primary Completion 2005-08 (Actual); Study Completion 2005-08 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Henning T Mouridsen, MD, Dr. med., Principal Investigator — Rigshospitalet, The Finsen Centre 5074, Blegdamsvej 9, DK-2100 Copenhagen
Locations (34):
- Denmark (15):
  - Aalborg Hospital South, Aalborg
  - Aarhus County Hospital, Aarhus
  - Aarhus Municipality Hospital, Aarhus
  - Rigshospitalet, Haematology Department, Copenhagen
  - Rigshospitalet, Oncology Department, Copenhagen
  - Esbjerg District Hospital, Esbjerg
  - Herlev County Hospital, Haematology Department, Herlev
  - Herlev County Hospital, Oncology Department, Herlev
  - Hilleroed Hospital, Hilleroed
  - Naestved District Hospital, Næstved
  - Odense University Hospital, Odense
  - Roskilde County Hospital, Roskilde
  - Soenderborg Hospital, Sønderborg
  - Vejle Hospital, Vejle
  - Viborg Hospital, Viborg
- Germany (9):
  - Evangelisches Bethesda Krankenhaus, Essen Borbak Statt
  - Klinik für Gynäkologie und Geburtshilfe, Frankfurt am Main
  - Klinik und Poliklinik für Innere Medizin, Hamburg
  - Medizinische Hochschule Hannover, Hanover
  - Universitäts Frauenklinik, Kiel
  - Universitäts Medizinische Klinik, Kiel
  - Frauenklinik com Roten Kreuz, Munich
  - Universitäts Frauenklinik, Rostock
  - Klinik für Gynäkologie und Gynäkologische Onkologie, Wiesbaden
- Italy (4):
  - Ospedale G.B. Morgagni L. Pierantoni, Forlì
  - Presidio Ospedaliero di Ravenna, Ravenna
  - Ospedale degli Infermi, Rimini
  - Ospedali Riuniti, Trieste
- Netherlands (3):
  - Willem Alexander Hospital, 's-Hertogenbosch
  - Netherland Cancer Institute, Amsterdam
  - University Hospital, Groningen
- Poland (3):
  - Centre of Oncology - Krakow Division, Krakow
  - Maria Sklodowska-Curie Memorial Cancer Center, Warsaw
  - Dolnoslaski Centrum Onkologii oddzial Chemoterapii, Wroclaw

REFERENCES:
- [Result] Mouridsen HT, Langer SW, Buter J, Eidtmann H, Rosti G, de Wit M, Knoblauch P, Rasmussen A, Dahlstrom K, Jensen PB, Giaccone G. Treatment of anthracycline extravasation with Savene (dexrazoxane): results from two prospective clinical multicentre studies. Ann Oncol. 2007 Mar;18(3):546-50. doi: 10.1093/annonc/mdl413. Epub 2006 Dec 21. PMID 17185744